CLINICAL TRIAL: NCT03540186
Title: A Nutritional Supplement Epigenome Antivir Combined With Acupuncture for the Treatment of Osteoarthritis Who Are Overweight or Obese
Brief Title: Epigenorm Antivir Combined With Acupuncture for the Treatment of Osteoarthritis Patients Who Are Overweight or Obese
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal State Budgetary Scientific Institution, Research Institute of Fundamental and Clinical Immunology (Other)
Responsible Party: Principal Investigator, Ivan Shirinsky, MD, PhD, Principal Investigator, Federal State Budgetary Scientific Institution, Research Institute of Fundamental and Clinical Immunology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCI002
Record Dates: First submitted 2018-05-08; First posted 2018-05-30 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Osteoarthritis; Overweight and Obesity
MeSH Terms: conditions — Osteoarthritis; Overweight; Obesity | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epigenorm Antivir and acupuncture arm (Experimental): Epigenorm Antivir is a dietary supplement containing extracts of glycyrrhiza roots, hippophae rhamnoides leaves, curcumin, green tea, and vitamin C. Acupuncture involves inserting needles at certain points of the body.
  Interventions: Dietary Supplement: Epigenorm Antivir; Procedure: Acupuncture

INTERVENTIONS:
Dietary Supplement: Epigenorm Antivir — 1 capsule of Epigenorm Antivir twice daily for 3 months
Procedure: Acupuncture — Acupuncture involves inserting sterile needles into the skin. The needles do not go into the skin very far. Number of acupuncture sessions: no less than 15 sessions, based on the physician discretion

SUMMARY:
The study evaluates analgesic, antiinflammatory and metabolic effects of a supplement Epigenome-Antivir (extracts of glycyrrhiza roots, hippophae rhamnoides leaves, curcumin, green tea, and vitamin C) combined with acupuncture in patients with knee osteoarthritis (OA) and metabolic syndrome.

DETAILED DESCRIPTION:
Epigenome-Antivir components have long been used in traditional medicine and have been shown to exert anti-inflammatory properties both in vitro and in vivo. It has also been shown that acupuncture can provide a moderate analgesic effect in osteoarthritis. It is anticipated that the combination of Epigenome-Antivir and acupuncture will reduce pain, inflammatory and metabolic markers in patients with OA and metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the knee fulfilling American College of Rheumatology (ACR) criteria
* BMI of 25 or more

Exclusion Criteria:

* use of NSAIDs one month prior to study entry (paracetamol is allowed)
* pregnancy and lactation
* increased sensitivity to the study drug
* clinically significant renal function impairment
* use of antidepressants
* diagnosis of bipolar disorder
* use of symptomatic slow acting drugs of OA (SYSADOA) one month prior to study entry
* any condition which may lead to difficulties to participation in the study from the viewpoint of Investigator

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-06-29 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Visual Analogue Scale for Pain | Baseline, 4 weeks, 8 weeks, 12 weeks
  The Visual Analogue Scale for Pain varies from 0 to 10 cm. Higher values represent worse outcomes.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) - subscale Pain | Baseline, 4 weeks, 8 weeks, 12 weeks
  KOOS Pain consists of 9 items, which are answered on a 4-point likert scale (0=no problems, 4=extreme problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee injury and Osteoarthritis Outcome Score (KOOS) - subscale Activities of daily living (ADL) | Baseline, 4 weeks, 8 weeks, 12 weeks
  KOOS ADL consists of 17 items, which are answered on a 4-point likert scale (0=no problems, 4=extreme problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee injury and Osteoarthritis Outcome Score (KOOS) - subscale Symptoms | Baseline, 4 weeks, 8 weeks, 12 weeks
  KOOS Symptoms consists of 7 items, which are answered on a 4-point likert scale (0=no problems, 4=extreme problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Quality of life with the The Short Form (36) Health Survey score | Baseline, 4 weeks, 8 weeks, 12 weeks
  he Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section.Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Intermittent and Constant Osteoarthritis Pain self-report questionnaire | Baseline, 4 weeks, 8 weeks, 12 weeks
  Pain measure: Scale range 0-100 with higher scores indicating worse pain
Changes in serum levels of aggrecan | Baseline, 8 weeks
  serum levels of aggrecan measured in ng/ml
Changes in serum levels of antibodies to collagen type II | Baseline, 8 weeks
  serum levels of antibodies to collagen type II measured AU/ml
Changes in serum levels of C-reactive protein | Baseline, 8 weeks
  serum levels of C-reactive protein (CRP), g/l
Changes in histamine levels | Baseline, 8 weeks
  serum levels of histamine in ng/ml
Changes in inflammation biomarkers | Baseline, 8 weeks
  serum levels of (CRP), interleukin (IL)-6, IL- 18, adiponectin, IL-10, and interferon (IFN) γ in pg/ml
Changes in lipid biomarkers | Baseline, 8 weeks
  serum total cholesterol, HDL, and LDL measured in mmol/L
Changes in depression scores measured with Patient Health Questionnaire-9 (PHQ9P) | Baseline, 4 weeks, 8 weeks, 12 weeks
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. It consists of nine questions with responses ranging from "0" (not at all) to "3" (nearly every day). The possible range is 0-27. Higher values represent worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Shirinsky, MD, PhD, Principal Investigator — Federal State Budgetary Scientific Institution, Research Institute of Fundamental and Clinical Immunology
Locations (1):
- Laboratory of Clinical Immunopharmacology, Novosibirsk, Russia